CLINICAL TRIAL: NCT01829542
Title: Dose-dependent Effects of Blueberry Polyphenols on Endothelial Function in Healthy Individuals
Acronym: BB2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Alpro Foundation (Other)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: BB2UReading
Record Dates: First submitted 2013-04-08; First posted 2013-04-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Endothelial Function
Keywords: flow-mediated dilation; blueberry polyphenols; dose-dependency
MeSH Terms: interventions — Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- 319 mg blueberry polyphenols (Active Comparator): Freeze-dried blueberry powder dissolved in water
  Interventions: Dietary Supplement: Freeze-dried blueberry powder dissolved in water
- 639 mg blueberry polyphenols (Active Comparator): Freeze-dried blueberry powder dissolved in water
  Interventions: Dietary Supplement: Freeze-dried blueberry powder dissolved in water
- 766 mg blueberry polyphenols (Active Comparator): Freeze-dried blueberry powder dissolved in water
  Interventions: Dietary Supplement: Freeze-dried blueberry powder dissolved in water
- 1466 mg blueberry polyphenols (Active Comparator): Freeze-dried blueberry powder dissolved in water
  Interventions: Dietary Supplement: Freeze-dried blueberry powder dissolved in water
- 1791 mg total blueberry polyphenols (Active Comparator): Freeze-dried blueberry powder dissolved in water
  Interventions: Dietary Supplement: Freeze-dried blueberry powder dissolved in water
- O mg blueberry polyphenols (Placebo Comparator): Macro- and micronutrient matched control drink
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Freeze-dried blueberry powder dissolved in water — Wild blueberry freeze-dried powder dissolved in water
  Arms: 1466 mg blueberry polyphenols; 1791 mg total blueberry polyphenols; 319 mg blueberry polyphenols; 639 mg blueberry polyphenols; 766 mg blueberry polyphenols
Dietary Supplement: Control — Macro- and micro-nutrient matched control in water
  Arms: O mg blueberry polyphenols

SUMMARY:
The purpose of this study is to assess the impact of acute blueberry polyphenol intake on endothelial function of healthy volunteers. Specifically, the investigators plan to perform a randomised, double blind, cross-over human intervention trial using a blueberry drink to investigate the dose-dependent effects of blueberry polyphenols on blood vessel function using Flow mediated dilation (FMD) to measure endothelial function. The study will not only measure the acute effects of flavonoid ingestion on vascular reactivity but will also assess plasma polyphenol metabolite levels.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-40 years
* Healthy
* signed consent form

Exclusion Criteria:

* Blood pressure > 140/90 mmHg
* Had suffered a myocardial infarction or stroke
* Suffers from any blood-clotting disorder
* Suffers from any metabolic disorders (e.g. diabetes or any other endocrine or liver diseases)
* Any dietary restrictions or on a weight reducing diet
* Allergies or intolerances to any foods
* Smoker
* Heavy drinker (>21 units per week)
* On any lipid-modifying medication
* On any blood pressure lowering medication
* On any medication affecting blood clotting
* Taking high dose fish oil supplements (greater then 1 g EPA and DHA per day) or high doses of antioxidant vitamins (greater then 800 μg vitamin A, 60 mg vitamin C, 10 mg vitamin E or 400 μg beta carotene)
* Taking probiotics, prebiotics, synbiotics, antibiotics or anti-inflammatory or blood lowering medication within a 2-month period prior to the study
* Planning on altering consumption of vitamin supplements/fish oil capsules during the course of the study
* Undertakes strenuous exercise > 4 times per week for > 1 hour per session
* Haemoglobin levels below reference range provided by the Royal Berkshire Hospital

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilation | 0-1 hour after consumption

SECONDARY OUTCOMES:
plasma blueberry polyphenol metabolites | 0-1 h after consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Hugh Sinclair Unit of Human Nutrition, Reading, Berkshire, United Kingdom

REFERENCES:
- [Derived] Rodriguez-Mateos A, Rendeiro C, Bergillos-Meca T, Tabatabaee S, George TW, Heiss C, Spencer JP. Intake and time dependence of blueberry flavonoid-induced improvements in vascular function: a randomized, controlled, double-blind, crossover intervention study with mechanistic insights into biological activity. Am J Clin Nutr. 2013 Nov;98(5):1179-91. doi: 10.3945/ajcn.113.066639. Epub 2013 Sep 4. PMID 24004888